CLINICAL TRIAL: NCT06815705
Title: An Exploratory Study of Reconstruction of Cervical Lymphatic System by Vascularized Lymphoid Tissue Transplantation During Head and Neck Squamous Cell Carcinoma Surgery
Brief Title: Reconstruction of Cervical Lymphatic System During Head and Neck Squamous Cell Carcinoma Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Youyuan Wang, Associate Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSJS-2024-074-02
Record Dates: First submitted 2024-12-23; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Lymphedema, Secondary; Neck Lymph Dissection; Vascularized Lymph Node Transplantation
Keywords: Vascularized lymph node transplantation; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascularized lymphatic transplantation (Experimental): Surgical methods According to the guidelines, the tumor was removed, the neck lymph node was removed, and the maxillofacial and neck defects were repaired with vascularized thoracic artery flap and axillary lymphatic tissue transplantation.
  Interventions: Procedure: Vascularized lymphatic transplantation

INTERVENTIONS:
Procedure: Vascularized lymphatic transplantation — Preoperative ultrasonography was performed to check the distribution, quantity and size of axillary lymph nodes. During the operation, methylene blue was injected subcutaneously into the elbow fossa to make the axillary lymph nodes in area B and D chromogenic, and avoid damage to the arm drainage lymph nodes.
  Adjusting the flap design according to the size of the defect. The perforating branches of lymphoid tissue in areas A and C of grade I were located about 3-5cm above the perforating branches of the skin, and moved towards the thoracic side to the lymphatic adipose tissue. Finally, the pedicle of the thoracic dorsal artery was separated, and the blood transport of the flap and the lymphatic adipose tissue was examined by fluorescence imaging and other methods. The lymphoid adipose tissue was placed in the neck area I and II, and fixed by suture. The arteriovenous microvessels in the thoracic dorsal were anastomosed to the vessels in the receiving area of neck.

SUMMARY:
Head and neck squamous cell carcinoma is one of the most common malignant tumors. At present, the standard treatment of head and neck squamous cell carcinoma recommended by the National Comprehensive Cancer Network(NCCN) treatment guideline in the United States and the Chinese Society of Clinical Oncology(CSCO) treatment guideline in China is a comprehensive treatment model based on surgery, supplemented by radiotherapy, chemotherapy, immunization and targeted therapy. Neck lymph dissection is one of the most important surgical procedures for the treatment of head and neck squamous cell carcinoma. The injury of surgery and postoperative adjuvant radiotherapy leads to inadequate drainage of lymphatic system, leading to head and neck lymphedema.

Vascularized lymph node transplantation is successfully used in the treatment of upper and lower limb lymphedema, but has not been reported in the treatment of head and neck lymphedema.

At present, neck lymph dissection is the standard surgical protocol for head and neck squamous cell carcinoma, and there is no clear evidence that neck lymph dissection can be avoided. The dorsal thoracic artery flap can be used to make the flap of chimeric axillary lymph node, and can also be used as one of the vascularized lymph transplantation donor areas for the treatment of lymphedema without increasing the risk of upper limb lymphedema in the donor area.

Therefore, the investigators propose: Can the function of the head and neck lymphatic system be reconstructed by transplanting normal lymph nodes from other parts of the body into the neck to form new lymphatic pathways at the same time of operation for head and neck squamous cell carcinoma? In our previous operation for head and neck squamous cell carcinoma, thoracic dorsal artery flap with partial axillary lymphoid tissue transplantation was used to repair head and neck defects. Retrospective analysis showed that the lymph node transplantation in the previous cases survived. Therefore, this project designed a prospective exploratory clinical study to clarify the activity and donor safety of cervical vascularized lymphatic transplantation, and further explore the effect of vascularized lymphatic tissue transplantation to rebuild the cervical lymphatic system in reducing the incidence of postoperative head and neck lymphedema, alleviating cervical fibrosis after radiotherapy and even improving the prognosis of patients.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma is one of the most common malignant tumors. At present, the standard treatment of head and neck squamous cell carcinoma recommended by the NCCN treatment guideline in the United States and the CSCO treatment guideline in China is a comprehensive treatment model based on surgery, supplemented by radiotherapy, chemotherapy, immunization and targeted therapy. Neck lymph dissection is one of the most important surgical procedures for the treatment of head and neck squamous cell carcinoma. The injury of surgery and postoperative adjuvant radiotherapy leads to inadequate drainage of lymphatic system, leading to head and neck lymphedema. Lymphedema is a progressive process that includes features such as lymphatic stasis, lymphatic vessel remodeling and dysfunction, inflammation, fatty tissue deposition, and eventually fibrosis. Therefore, in addition to edema, complications such as cervical fibrosis may occur, which seriously affects the quality of life of patients with head and neck squamous cell carcinoma. In addition, the absence of lymphatic tissue in the neck after cervical lymph dissection may damage the local lymphatic immune monitoring function of the head and neck, and affect the postoperative therapeutic effect and prognosis of patients.

Surgical treatment of head and neck lymphedema includes lymphatic venous shunt and vascularized lymph node transplantation, which involves the transfer of healthy lymph nodes from unaffected parts of the body to the site of lymphedema. Vascularized lymph node transplantation is successfully used in the treatment of upper and lower limb lymphedema, but has not been reported in the treatment of head and neck lymphedema.

At present, neck lymph dissection is the standard surgical protocol for head and neck squamous cell carcinoma, and there is no clear evidence that neck lymph dissection can be avoided. Therefore, head and neck lymphedema after head and neck squamous cell carcinoma is a common surgical complication. In our previous study, the investigators collected the data of 71 patients with head and neck squamous cell carcinoma undergoing surgical treatment, and found that the greater the scope of cervical lymph dissection, the more serious the degree of lymphedema after surgery. In addition, our research group has successfully implemented thoracic dorsal artery flap to repair oral cancer defects in more than 100 cases in the early stage, which proved that the success rate of thoracic dorsal artery flap is high and the functional injury of the donor area is small. The dorsal thoracic artery flap can be used to make the flap of chimeric axillary lymph node, and can also be used as one of the vascularized lymph transplantation donor areas for the treatment of lymphedema without increasing the risk of upper limb lymphedema in the donor area.

There are no effective preventive measures for head and neck lymphedema and neck fibrosis in patients with head and neck squamous cell carcinoma after comprehensive treatment. In order to reduce the pain, cost and possibility of reoperation caused by postoperative treatment, the prevention of head and neck lymphedema after the operation of head and neck squamous cell carcinoma has become an important clinical problem to be solved in this project. Therefore, the investigators propose: Can normal lymph nodes from other parts of the body be transplanted into the neck to form new lymphatic pathways during head and neck squamous cell carcinoma surgery to rebuild the function of the head and neck lymphatic system and avoid postoperative complications such as lymphedema? In our previous study, 6 patients with head and neck squamous cell carcinoma were successfully transplanted with dorsal thoracic artery flap carrying part of armpit lymphoid tissue during operation to reconstruct the neck lymphatic system. Postoperative Magnetic Resonance(MR) And ultrasound showed that the size and structure of the transplanted lymph nodes were normal, no lymph node necrosis was observed, and blood flow was lymphatic portal type. No upper limb lymphedema occurred in the donor area.

In this study, patients with head and neck squamous cell carcinoma with clinical stages of T2-3,N0-3,M0 and T4a,N0-3,M0 requiring surgical treatment and repair by skin flap transplantation were selected, and were enrolled by Simon stage II, and the intervention measures were based on the recommended surgical methods in the guidelines and the vascularization axillary lymphatic transplantation at the same time. The main study endpoints were the survival of transplanted lymph nodes, the incidence and degree of lymphedema in the head and neck, and the incidence and degree of lymphedema in the upper limb of the donor area. Secondary endpoints were 2-year disease-free survival, 2-year overall survival, patient quality of life evaluation, and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. This study selected T2-3,N0-3,M0; Patients with T4a,N0-3,M0 head and neck squamous cell carcinoma (AJCC 8th) can be treated surgically with flap repair and no axillary lymphatic metastasis.
2. No history of other malignant tumors 3.18-75 years old

4. Baseline check is normal:

1. In the past 14 days without the use of granulocyte colony-stimulating factor, the absolute value of neutrophil (ANC) ≥1.5x109/L;
2. Platelets ≥100×109/L in the past 14 days without blood transfusion;
3. Hemoglobin >9g/dL in the last 14 days without blood transfusion or use of erythropoietin;
4. Total bilirubin ≤1.5× upper limit of normal (ULN);
5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft- Gault formula) ≥60 ml/min;
7. Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
9. The myocardial enzyme profile is within the normal range (if the researchers comprehensively judge that the simple laboratory abnormality is not clinically significant, it is also allowed to be included);
10. For female subjects of reproductive age, a urine or serum pregnancy test should be taken and the result is negative within 3 days prior to the first treatment (day

    1 of cycle 1). If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
11. If there is a risk of conception, all subjects (male or female) should use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last treatment (or 180 days after the last chemotherapy drug administration).
12. No axillary lymph node metastasis.

Exclusion Criteria:

1. Diagnosis of other malignant tumors, or treatment of HNSCC did not start.
2. Prior to treatment, an active autoimmune disease requiring systemic treatment (e.g. use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within the previous 2 years. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
3. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
4. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
5. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the research center);

   Note: Hepatitis B subjects who meet the following criteria can also be enrolled:
   1. Pre-treatment HBV viral load <1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy throughout study treatment to avoid viral reactivation
   2. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required
6. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
7. Pregnant or lactating women;
8. The presence of any serious or uncontrolled systemic disease, such as:

   1. The resting electrocardiogram has major abnormal rhythm, conduction or morphology, such as complete left bundle branch block, heart block above Ⅱ degree, ventricular arrhythmia or atrial fibrillation;
   2. Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure;
   3. Any arterial thrombosis, embolism or ischemia occurred within 6 months before treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack;
   4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
   5. There is a history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to treatment, or there is currently clinically active interstitial lung disease;
   6. Active pulmonary tuberculosis;
   7. There is an active or uncontrolled infection that requires systemic treatment;
   8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
   9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
   10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
   11. Urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0 g;
   12. Patients with mental disorders who cannot cooperate with treatment;
9. Axillary lymphatic metastasis
10. Medical history or evidence of disease that may interfere with the test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of head and neck lymphedema within 2 years after surgery | At least 3 months to 2 years after surgery
  Head and neck lymphedema refers to external and internal head and neck lymphedema caused by disruption of lymphatic pathways due to surgical neck lymph node dissection or radiotherapy. This disruption prevents lymphatic fluid from flowing from the soft tissue interstitium of the head and neck to the right lymphatic vessel and the left thoracic duct. The incidence rate of head and neck lymphedema within 2 years refers to the proportion of patients with head and neck lymphedema from at least 3 months to 2 years after surgery in all patients who underwent vascularized lymphatic transplantation. The degree of head and neck lymphedema is divided into 5 grades according to the MD Anderson Cancer Center(MDACC) Head and neck lymphedema(HNL) rating scale.
severity of head and neck lymphedema within 2 years after surgery | At least 3 months to 2 years after surgery
  The degree of lymphedema was determined by comparing MRI images before and after treatment, and the thickness of the most severely affected area increased by no more than 50% compared with the original thickness, which was mild lymphedema. When the thickness increases between 50% and 100%, it is moderate lymphedema. When the thickness increases by more than 100%, it is severe lymphedema.

SECONDARY OUTCOMES:
The survival of transplanted lymph nodes at 3 months and 6 months after comprehensive treatment | 3，6，12，24 months after comprehensive treatment
  The number, morphology and hemodynamics of transplanted lymph nodes at 3, 6, 12 and 24 months after treatment were measured by color Doppler ultrasound, magnetic resonance imaging and radionuclide lymphography. Ultrasound showed that the blood flow signal of the surviving transplanted lymph nodes was lymphatic portal type.
Incidence of upper limb lymphedema in donor area | At least 6 months to 2 years after surgery
  The proportion of patients with upper limb lymphedema at the donor site from at least 6 months to 2 years after surgery in all patients who were repaired with vascularized lymphedema free thoracic dorsal artery flap. The diagnosis of upper limb lymphedema was referred to a prospective clinical study conducted by the Mayo Clinic in the United States, in which bilateral upper limb circumference was measured every 5cm from the wrist transverse line to the axillary line. The edema volume used was defined as a postoperative interlimb difference of ≥10% from baseline. The formula was used to calculate the volume change: [([VIp-VIb] / Vib) 100]-[([Vcp-Vcb] / Vcb) 100%], where Vip is the volume of the postoperative arm on the same side; Vib is the baseline volume of the ipsilateral arm; Vcp is the volume of the contralateral arm after surgery; The Vcb is the baseline volume of the opposite arm at baseline.
degree of upper limb lymphedema in donor area | At least 6 months to 2 years after surgery
  The degree of edema was evaluated using the World Health Organization lymphedema staging method, upper limb arm circumference measurement, shoulder joint range of motion, and ultrasonic measurement of skin and subcutaneous tissue thickness.
2-year disease-free survival | within 2 years after surgery
  Proportion of patients who did not have disease recurrence or death within 2 years after receiving standard surgery in this program.
2-year overall survival | within 2 years after surgery
  Proportion of patients who did not die from any cause within 2 years of receiving standard surgery.
Postoperative magnetic resonance lymphangiography was performed by injecting contrast agent into the flap to check the number of transplanted lymph nodes | 3，6，12，24 months after comprehensive treatment
  Preoperative and postoperative magnetic resonance lymphangiography was performed by subcutaneous injection of contrast agent to detect the difference of lymphatic network connectivity in the lymphatic tissue before and after transplantation, and to detect whether the transplanted lymph nodes formed a new lymphatic network with the remaining lymphatic tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Youyuan, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
We use EDC data repositories where other researchers can access it. The sharing of IPD must typically be approved by an ethics committee or institutional review board (IRB) to ensure compliance with privacy laws and regulations (such as HIPAA in the U.S., GDPR in the EU, etc.). We alos set up a committee to oversee the sharing of IPD, ensuring that the data is used responsibly and in accordance with ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the primary study results are published, within 5 years after the study is published
Access Criteria: 1. Access is typically granted only to researchers with legitimate scientific or public health research aims.
     Researchers must usually provide evidence that their proposed study has been approved by an Institutional Review Board or Ethics Committee.
  2. The precise research purpose for which the IPD can be used, and not for unrelated or commercial purposes.
     Researchers required to properly acknowledge the original study team in any publications or presentations based on the data.
  3. Access is granted with the expectation that the researcher will ensure participant privacy is maintained.
     Researchers must comply with relevant data protection laws.
  4. IPD may only be used for specific types of secondary research, such as exploratory analyses, meta-analyses, or validation studies. No Commercial Exploitation.
  5. We may require periodic reporting or auditing to ensure that the data is being use.

REFERENCES:
- [Background] Cohen O, Brauer PR, Judson BL, Burtness BA, Earles J, Mehra S. Guideline - Adherence in advanced stage head and neck cancer is associated with improved survival - A National study. Oral Oncol. 2022 Feb;125:105694. doi: 10.1016/j.oraloncology.2021.105694. Epub 2021 Dec 28. PMID 34971883
- [Background] Vos JL, Elbers JBW, Krijgsman O, Traets JJH, Qiao X, van der Leun AM, Lubeck Y, Seignette IM, Smit LA, Willems SM, van den Brekel MWM, Dirven R, Baris Karakullukcu M, Karssemakers L, Klop WMC, Lohuis PJFM, Schreuder WH, Smeele LE, van der Velden LA, Bing Tan I, Onderwater S, Jasperse B, Vogel WV, Al-Mamgani A, Keijser A, van der Noort V, Broeks A, Hooijberg E, Peeper DS, Schumacher TN, Blank CU, de Boer JP, Haanen JBAG, Zuur CL. Neoadjuvant immunotherapy with nivolumab and ipilimumab induces major pathological responses in patients with head and neck squamous cell carcinoma. Nat Commun. 2021 Dec 22;12(1):7348. doi: 10.1038/s41467-021-26472-9. PMID 34937871
- [Background] Savvides PP. The role of chemotherapy in the management of patients with head and neck cancer. Semin Plast Surg. 2010 May;24(2):137-47. doi: 10.1055/s-0030-1255331. PMID 22550434
- [Background] Deng J, Ridner SH, Dietrich MS, Wells N, Wallston KA, Sinard RJ, Cmelak AJ, Murphy BA. Prevalence of secondary lymphedema in patients with head and neck cancer. J Pain Symptom Manage. 2012 Feb;43(2):244-52. doi: 10.1016/j.jpainsymman.2011.03.019. Epub 2011 Jul 30. PMID 21802897
- [Background] Stubblefield MD, Weycker D. Under recognition and treatment of lymphedema in head and neck cancer survivors - a database study. Support Care Cancer. 2023 Mar 23;31(4):229. doi: 10.1007/s00520-023-07698-3. PMID 36952136
- [Background] Deng J, Lukens JN, Swisher-McClure S, Cohn JC, Spinelli BA, Quinn RJ, Chittams J, McMenamin E, Lin A. Photobiomodulation Therapy in Head and Neck Cancer-Related Lymphedema: A Pilot Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211037938. doi: 10.1177/15347354211037938. PMID 34387119
- [Background] Schaverien MV, Asaad M, Selber JC, Liu J, Chen DN, Hall MS, Butler CE. Outcomes of Vascularized Lymph Node Transplantation for Treatment of Lymphedema. J Am Coll Surg. 2021 Jun;232(6):982-994. doi: 10.1016/j.jamcollsurg.2021.03.002. Epub 2021 Mar 22. PMID 33766726
- [Background] Coroneos CJ, Asaad M, Wong FC, Hall MS, Chen DN, Hanasono MM, Schaverien MV. Outcomes and technical modifications of vascularized lymph node transplantation from the lateral thoracic region for treatment of lymphedema. J Surg Oncol. 2022 Mar;125(4):603-614. doi: 10.1002/jso.26783. Epub 2022 Jan 6. PMID 34989418
- [Background] Poon Y, Wei CY. Vascularized groin lymph node flap transfer for postmastectomy upper limb lymphedema: flap anatomy, recipient sites, and outcomes. Plast Reconstr Surg. 2014 Mar;133(3):428e. doi: 10.1097/01.prs.0000438451.45227.b6. No abstract available. PMID 24572896
- [Background] Deng H, Zhou J, Chen H, Cai X, Zhong R, Li F, Cheng B, Li C, Jia Q, Zhou C, Petersen RH, Rocco G, Brunelli A, Ng CSH, D'Amico TA, Su C, He J, Liang W, Zhu B; AME Thoracic Surgery Collaborative Group. Impact of lymphadenectomy extent on immunotherapy efficacy in postresectional recurred non-small cell lung cancer: a multi-institutional retrospective cohort study. Int J Surg. 2024 Jan 1;110(1):238-252. doi: 10.1097/JS9.0000000000000774. PMID 37755384
- [Background] Fear VS, Forbes CA, Neeve SA, Fisher SA, Chee J, Waithman J, Ma SK, Lake R, Nowak AK, Creaney J, Brown MD, Saunders C, Robinson BWS. Tumour draining lymph node-generated CD8 T cells play a role in controlling lung metastases after a primary tumour is removed but not when adjuvant immunotherapy is used. Cancer Immunol Immunother. 2021 Nov;70(11):3249-3258. doi: 10.1007/s00262-021-02934-3. Epub 2021 Apr 9. PMID 33835222
- [Background] Rahim MK, Okholm TLH, Jones KB, McCarthy EE, Liu CC, Yee JL, Tamaki SJ, Marquez DM, Tenvooren I, Wai K, Cheung A, Davidson BR, Johri V, Samad B, O'Gorman WE, Krummel MF, van Zante A, Combes AJ, Angelo M, Fong L, Algazi AP, Ha P, Spitzer MH. Dynamic CD8+ T cell responses to cancer immunotherapy in human regional lymph nodes are disrupted in metastatic lymph nodes. Cell. 2023 Mar 16;186(6):1127-1143.e18. doi: 10.1016/j.cell.2023.02.021. PMID 36931243
- [Background] Huang Q, Wu X, Wang Z, Chen X, Wang L, Lu Y, Xiong D, Liu Q, Tian Y, Lin H, Guo J, Wen S, Dong W, Yang X, Yuan Y, Yue Z, Lei S, Wu Q, Ran L, Xie L, Wang Y, Gao L, Tian Q, Zhou X, Sun B, Xu L, Tang Z, Ye L. The primordial differentiation of tumor-specific memory CD8+ T cells as bona fide responders to PD-1/PD-L1 blockade in draining lymph nodes. Cell. 2022 Oct 27;185(22):4049-4066.e25. doi: 10.1016/j.cell.2022.09.020. Epub 2022 Oct 7. PMID 36208623

DOCUMENTS (1):
  • Informed Consent Form (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT06815705/ICF_000.pdf